CLINICAL TRIAL: NCT06235827
Title: Effects of Green Tea Consumption on Retinal Nerve Fiber Layer ( RNFL) and Intraocular Pressure ( IOP) in Patients With Primary Glaucoma
Brief Title: Effects of Green Tea Consumption on Primary Glaucoma
Acronym: GTG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Siti Sarah Binti Shokri, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RSCH ID-23-03868-NIT
Record Dates: First submitted 2023-10-06; First posted 2024-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Primary Glaucoma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green tea group (Experimental): Patients in Group A will have to consume two cup (250ml for each cup) of hot green tea, five days per week for 6 months. A tea bag is brewed in 250ml hot water for 3 minutes.
  Interventions: Dietary Supplement: Green tean group
- Control Group (Experimental): Patients in Group B will not consume green tea for 6 months during study period.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Green tean group — Patients in Group A will have to consume two cups (250ml for each cup) of hot green tea, five days per week for 6 months. A tea bag is brewed in 250ml hot water for 3 minutes. They are only allowed to consume as hot drink, not for iced tea. Any sweetener or sugar is not allowed to mix in the drink. The green tea bag will be distributed to patient at beginning of research and at every visit. Patient will be reminded weekly using text messages or phone call by a research assistant for green tea consumption.
  Arms: Green tea group
Dietary Supplement: Control group — Patients in Group B will not be consuming green tea during 6 months of study period.
  Arms: Control Group

SUMMARY:
The goal of this randomised control trial is to learn about the effect of green tea consumption on patients with primary glaucoma.

The main questions to answer are:

1. Is there any difference of intraocular pressure (IOP) in patient with primary glaucoma after 1 month, 3 months and 6 months who is consuming green tea compared to patient not consuming green tea?
2. Is there any difference of retina nerve fibre layer in patient with primary glaucoma after 1 month, 3months and 6 months who is consuming green tea compared to patient not consuming green tea?

Researchers will compare patients with primary glaucoma who are consuming green tea and normal daily drinking to see if any affect to intraocular pressure and retina nerve fibre layer.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy characterised by loss of retinal ganglion cells (RGCs) with corresponding visual field loss. The current established treatment of glaucoma is by reducing IOP, as one of neuroprotectant factor to prevent further loss RGCs. However, it is not always sufficient to fully prevent disease progression. Oxidative stress is one of biological insult contribute to etiology and progression of glaucoma. Antioxidants represent the first line of defence against oxidative stress and are obtained through the diet and produced internally has shown to be protective towards glaucoma. Green tea is one of the most antioxidant rich drink due to its high content of flavonoids commonly known as catechins.

The investigator would like to evaluate the effect of 6 months consumption of green tea on intraocular pressure (IOP) and retinal nerve fibre layer thickness (RNFL) in patients with primary glaucoma. This is a randomised controlled study involving primary glaucoma patients who are attending ophthalmology clinic at Hospital Universiti Sains Malaysia. Evaluation of study sample includes baseline ocular examination, IOP and Optical Coherence Tomography Retinal Nerve Fibre Layer (OCT RNFL). Subjects who fulfil the inclusion and exclusion criteria for the study will be selected.

Patients in Group A will consume two cups per day (250ml for each cup) of hot green tea, five days per week for 6 months while other Group B (control group) will not consume green tea. IOP and OCT RNFL measurement will be taken at baseline, first month, 3rd month and 6th month post recruitment of subjects. All patients will be given dietary diary to note down their daily drinks' consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of primary glaucoma (POAG/PACG/NTG) that achieve target IOP with medical therapy at least for 6 months.
* Never consume green tea as daily drinks.

Exclusion Criteria:

* Dense cataract with Lens Opacity Classification Sytem (LOCS II) of more than grade 2
* Any other ocular media opacity that may interfere with OCT imaging ( eg: cornea scar/vitreous haemorrhage)
* Any history of optic neuropathy
* History of glaucoma or retinal surgery
* Macular degeneration and retinal disorder
* Patient with caffein sensitive that causes unpleasant reaction (eg: palpitation, insomnia, nausea, constipation)
* Allergic to green tea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effect of green tea consumption on intraocular pressure in patient with primary glaucoma | IOP measurement will be taken at baseline, first, and 6th-month post recruitment for group A and B.
  IOP measurement will be done using Goldmann Applanation Tonometer (GAT) for group A and Group B
Effect of green tea consumption on retinal nerve fiber layer thickness ( RNFL) in patient with primary glaucoma | OCT RNFL will be conducted at baseline, 1 month, 3 month and 6 month post recruitment for group A and B.
  Spectral domain Heidelberg Spectralis OCT will be used to measure RNFL thickness

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Siti Sarah Shokri, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braakhuis A, Raman R, Vaghefi E. The Association between Dietary Intake of Antioxidants and Ocular Disease. Diseases. 2017 Jan 30;5(1):3. doi: 10.3390/diseases5010003. PMID 28933356
- [Background] Chu KO, Chan KP, Wang CC, Chu CY, Li WY, Choy KW, Rogers MS, Pang CP. Green tea catechins and their oxidative protection in the rat eye. J Agric Food Chem. 2010 Feb 10;58(3):1523-34. doi: 10.1021/jf9032602. PMID 20085274
- [Background] Henning SM, Fajardo-Lira C, Lee HW, Youssefian AA, Go VL, Heber D. Catechin content of 18 teas and a green tea extract supplement correlates with the antioxidant capacity. Nutr Cancer. 2003;45(2):226-35. doi: 10.1207/S15327914NC4502_13. PMID 12881018
- [Background] Hu J, Webster D, Cao J, Shao A. The safety of green tea and green tea extract consumption in adults - Results of a systematic review. Regul Toxicol Pharmacol. 2018 Jun;95:412-433. doi: 10.1016/j.yrtph.2018.03.019. Epub 2018 Mar 24. PMID 29580974
- [Background] Chen JZ, Kadlubar FF. A new clue to glaucoma pathogenesis. Am J Med. 2003 Jun 1;114(8):697-8. doi: 10.1016/s0002-9343(03)00199-2. No abstract available. PMID 12798460
- [Background] Kang JH, Ivey KL, Boumenna T, Rosner B, Wiggs JL, Pasquale LR. Prospective study of flavonoid intake and risk of primary open-angle glaucoma. Acta Ophthalmol. 2018 Sep;96(6):e692-e700. doi: 10.1111/aos.13705. Epub 2018 Mar 14. PMID 29536641
- [Background] Calandrella N, De Seta C, Scarsella G, Risuleo G. Carnitine reduces the lipoperoxidative damage of the membrane and apoptosis after induction of cell stress in experimental glaucoma. Cell Death Dis. 2010 Aug 5;1(8):e62. doi: 10.1038/cddis.2010.40. PMID 21364667
- [Background] Mousa A, Kondkar AA, Al-Obeidan SA, Azad TA, Sultan T, Osman E, Abu-Amero KK. Association of total antioxidants level with glaucoma type and severity. Saudi Med J. 2015 Jun;36(6):671-7. doi: 10.15537/smj.2015.6.10697. PMID 25987108
- [Background] Yang Y, Xu C, Chen Y, Liang JJ, Xu Y, Chen SL, Huang S, Yang Q, Cen LP, Pang CP, Sun XH, Ng TK. Green Tea Extract Ameliorates Ischemia-Induced Retinal Ganglion Cell Degeneration in Rats. Oxid Med Cell Longev. 2019 Jul 9;2019:8407206. doi: 10.1155/2019/8407206. eCollection 2019. PMID 31379990
- [Background] Falsini B, Marangoni D, Salgarello T, Stifano G, Montrone L, Di Landro S, Guccione L, Balestrazzi E, Colotto A. Effect of epigallocatechin-gallate on inner retinal function in ocular hypertension and glaucoma: a short-term study by pattern electroretinogram. Graefes Arch Clin Exp Ophthalmol. 2009 Sep;247(9):1223-33. doi: 10.1007/s00417-009-1064-z. Epub 2009 Mar 17. PMID 19290537
- [Background] Gasiunas K, Galgauskas S. Green tea-a new perspective of glaucoma prevention. Int J Ophthalmol. 2022 May 18;15(5):747-752. doi: 10.18240/ijo.2022.05.09. eCollection 2022. PMID 35601179
- [Background] Bernatoniene J, Kopustinskiene DM. The Role of Catechins in Cellular Responses to Oxidative Stress. Molecules. 2018 Apr 20;23(4):965. doi: 10.3390/molecules23040965. PMID 29677167

DOCUMENTS (1):
  • Study Protocol (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT06235827/Prot_000.pdf